CLINICAL TRIAL: NCT05043025
Title: Comparison of Patient Positions for Locating the Cricothyroid Membrane
Brief Title: Patient Positions for Locating the Cricothyroid Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 08-2021
Record Dates: First submitted 2021-08-31; First posted 2021-09-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cricothyroid Membrane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck extension group (Active Comparator): The cricothyroid membrane is identified in a neck extended position.
  Interventions: Other: Identification of the cricothyroid membrane
- Modified ramped position group (Experimental): The cricothyroid membrane is identified in a modified ramped position.
  Interventions: Other: Identification of the cricothyroid membrane

INTERVENTIONS:
Other: Identification of the cricothyroid membrane — The cricothyroid membrane is identified using a laryngeal handshake technique in different patient positions.

SUMMARY:
Cricothyroidotomy is an emergency rescue technique to secure the airway in a 'Can't intubate, Can't Oxygenate' (CICO) situation. The cricothyroid membrane (CTM) is the target site of cricothyroidotomy, and accurate identification of the CTM is essential for successful cricothyroidotomy. In this study, the investigators compare patient positions (neck extension vs. modified ramped position) in terms of the success rate for identifying the CTM in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* body mass index >30 kg/m2

Exclusion Criteria:

* anatomical abnormalities or pathologies of the neck
* a history of neck surgery
* cervical spine disorders
* skin lesions on the neck

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Success rate for the correct identification of the cricothyroid membrane | Immediately after identifying the cricothyroid membrane using a laryngeal handshake technique
  After identifying the cricothyroid membrane using a laryngeal handshake technique in different head positions, an assessor evaluates the correctness of its localization using ultrasound.

SECONDARY OUTCOMES:
Duration for identifying the cricothyroid membrane | At 90 seconds after administering neuromuscular blockade
  Time taken to locate the cricothyroid membrane is checked.
Distances between the center of the actual and perceived cricothyroid membrane | Immediately after identifying the cricothyroid membrane using a laryngeal handshake technique
  Distances between the center of the actual and perceived cricothyroid membrane is measured using ultrasound.
Perceived difficulty during cricothyroid membrane identification | At 5 minutes after identifying the cricothyroid membrane using a laryngeal handshake technique
  Anatomical difficulty perceived by the anesthesiologists during cricothyroid membrane identification is assessed (1, very easy; 2, easy; 3, moderate; 4, difficult; and 5, very difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Select State/Province, South Korea